CLINICAL TRIAL: NCT05773417
Title: Changes in Quality of Recovery With Low-Flow Anesthesia in Minor ENT Surgery (QoRLowflow)
Brief Title: Changes in Quality of Recovery With Low-Flow Anesthesia (QoRinLowflow)
Acronym: (QoRLowflow
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Acibadem University (Other)
Collaborators: Ataturk University (Other)
Responsible Party: Sponsor
Other Study IDs: Recovery quality 2122
Record Dates: First submitted 2023-01-18; First posted 2023-03-17 (Actual); Last update posted 2023-03-17 (Actual); Status verified 2023-03

CONDITIONS: Low Flow Anesthesia
Keywords: Low Flow Anesthesia; Quality of Recovery; Cognition Tests; Postoperative Complications
MeSH Terms: conditions — Postoperative Complications

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Low Flow: 0.5 L/minute
- High Flow: 4 L/minute

SUMMARY:
Postoperative recovery quality is as important as patient satisfaction and clinical results in terms of a fast and high-quality surgical process. This study was conducted to investigate the effect of low-flow anesthesia applications on the quality of patient recovery by evaluating the 'Quality of Recovery' (QoR40) test and the perception tests (PQRS Cognitive test) performed in the early postoperative period.

DETAILED DESCRIPTION:
All patients will be evaluated preoperatively in the anesthesia outpatient clinic, their consent will be obtained, and they will be informed about the 'Postoperative Recovery Evaluation' and pre-tests will be performed. All patients will receive premedication midazolam 0.07mg/kg intramuscularly 20 minutes before the operation. In both groups, anesthesia induction will be achieved with intravenous propofol 3 mg/kg, remifentanil 0.1 mic/kg, and rocuronium 0.06 mg/kg. Following endotracheal intubation, maintenance of anesthesia will be provided to the patients in Group I by inhalation, with sevoflurane MAC 1 in O2/Air 1/3 (4lt/min). On the other hand, patients in Group II will be switched to O2/Air 0.16/0.48 (0.5 lt/min) low flow anesthesia 15 minutes after the depth of anesthesia is provided (BIS<50) and inhalation anesthesia starts. Remifentanil infusion will be administered intravenously at 0.025-0.1 mic/kg/min to all patients in both groups for peroperative analgesia. For postoperative analgesia, fentanyl will be administered intravenously as 2 mic/kg 10 minutes before the end of the surgery. In group I patients, remifentanil infusion and inhalation anesthesia will be reduced and stopped at the end of surgery. (BIS maximum 60). In patients in Group II, inhalation anesthesia will be terminated 15 minutes before the end of surgery, and remifentanil infusion will be terminated with the last suture. (BIS maximum 60). Peroperatively, patients' heart rate, mean blood pressure, oxygen saturation with pulse oximetry, tidal volume, respiratory rate, inspiratory/expiratory oxygen/air/sevoflurane concentrations, leakage amounts, end tidal CO2 and inspiratory CO2 amounts, BIS values will be recorded at 15-minute intervals. . The end of the surgery, the last suture of the surgery, the end of the anesthesia will be recorded as the termination of the administration of intravenous and inhalation anesthetics. Muscle laxity of the patients will be restored with sugammadex 2 mg/kg. As the extubation criteria, the spontaneous ventilation of the patients with sufficient tidal volume and the end of muscle relaxation will be taken as BIS >70. The extubation time will be recorded. Postoperative recovery evaluations of the patients will be made. Nausea/vomiting and Modified Aldrete scores and VAS values of the patients followed for 30 minutes in the recovery unit will be recorded. At the end of the first 30 minutes, PQRS Cognitive test will be applied to the patients. On the morning of the first postoperative day, the QoR40 test will be applied and scored by an anesthesia technician who does not know the anesthesia method. The results will be compared.

ELIGIBILITY:
Inclusion Criteria:

1. Cases in which general anesthesia will be applied by intubation and anesthesia will be maintained with inhalation anesthetics;
2. 2 - 6 hour cases
3. 18 - 60 years old
4. Low flow anesthesia application with 0.5 lt/min flow rate
5. Patients undergoing muscular recovery with sugammadex

Exclusion Criteria:

1. Patients with bleeding diathesis or patients with bleeding in excess of 400 ml
2. Patients with mental/neurological problems
3. Patients who refused to participate in the study and could not respond
4. Patients who cannot apply low current
5. Uncooperative patients with delirium
6. Hypotension in perioperative parameters (MAP < 40 mmHg)
7. Patients with diabetic ketoacidosis
8. Cases taken when soda lime is dry

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Tertiary Care Clinic
Sampling Method: Probability Sample
Enrollment: 50 (Estimated)
Dates: Start 2021-01-01 (Actual); Primary Completion 2023-04-29 (Estimated); Study Completion 2023-05-01 (Estimated)

PRIMARY OUTCOMES:
The effect of low-flow anesthesia applications on the quality of patient recovery by evaluating the 'Quality of Recovery' performed in the early postoperative period. | Up to 2 days
  This questionnaire consists of 40 questions with 5 different aspects; emotional state (9 questions), physical comfort (12 questions), psychological support (7 questions), physical independence (5 questions), pain (7 questions). Each question will be answered as 'never', 'sometimes', 'often', 'often', 'always' according to the Likert scale, according to the frequency of occurrence. Each frequency term will be scored from 1 to 5.
  The questionnaire has parts A and B. In part A, the questions indicate positive aspects, the higher the frequency of occurrence, the higher the score. In part B, the opposite is true. In Part A, 'never' is denoted by '1', 'sometimes' by '2', often' by 3, often' by '4', 'always' by '5' . In part B, 'never' is expressed with '5', sometimes', '4', and so on. The total score ranges from QoR-40 40 (poor compilation) to 200 points (excellent compilation).

CONTACTS AND LOCATIONS:
Overall Officials: Serpil Z Ustalar, doctor, Principal Investigator — Acıbadem Mehmet Ali Aydınlar University
Locations (1):
- Acıbadem Mehmet Ali Aydınlar University, Istanbul, Üsküdar, Turkey (Türkiye)

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Result] Royse CF, Newman S, Chung F, Stygall J, McKay RE, Boldt J, Servin FS, Hurtado I, Hannallah R, Yu B, Wilkinson DJ. Development and feasibility of a scale to assess postoperative recovery: the post-operative quality recovery scale. Anesthesiology. 2010 Oct;113(4):892-905. doi: 10.1097/ALN.0b013e3181d960a9. PMID 20601860
- [Result] Jakobsson J. Assessing recovery after ambulatory anaesthesia, measures of resumption of activities of daily living. Curr Opin Anaesthesiol. 2011 Dec;24(6):601-4. doi: 10.1097/ACO.0b013e32834c3916. PMID 21945921